CLINICAL TRIAL: NCT00471302
Title: Establishment of Normal Immunological Parameters Among Healthy Volunteers in Kambila, Tieneguebougou, and Kalifabougou, Mali
Brief Title: Normal Immunological Parameters Among Healthy Volunteers in Kambila, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Bamako (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907141; 07-I-N141
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Malaria
Keywords: Immunology; Mali; Donor; Natural History
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy adults in a malaria endemic area in Mali

SUMMARY:
This study will determine the immune response to malaria infection in healthy volunteers compared with malaria patients. Malaria affects millions of people in Mali and Africa. It can cause fever, headaches, body aches, and weakness. Without treatment, the disease can be very serious in children. Developing an effective vaccine against the parasite that causes malaria is a crucial step toward controlling the disease; however, vaccines tested so far have provided very short-lived protection. A better understanding of the natural immunity to malaria may provide insight that can be applied to developing a more effective vaccine.

People 18 years of age or older who live in Kambila, Tieneguebougou or Kalifabougou, Mali, and are in good health may be eligible for this study.

Participants undergo a complete physical examination at the start of the study and then once a year for the 4-year duration of the study. They have a maximum of nine clinic visits a year to collect blood samples for research. The visits last about one hour, including a 30-minute observation time after the blood draw.

DETAILED DESCRIPTION:
Malaria results in at least 2.7 million deaths per year, the majority among African children. The development of a vaccine

against Plasmodium falciparum is regarded as a crucial step toward control of this disease. Unfortunately, vaccine

candidates have resulted in short-lived protection at best. The ineffectiveness of current vaccines may reflect the kinetics

of naturally acquired immunity to malaria in that multiple infections are required over years before partial protection is

achieved and then immunity is lost, or becomes less effective, in the absence of recurrent infection. The mechanisms

underlying the delayed acquisition and presumably rapid loss of humoral immunity are poorly understood. A more

detailed understanding of these processes at the cellular level may be important for vaccine development. We are

currently studying the cellular basis of humoral immunity to P. falciparum through research collaboration between the

Malaria Research and Training Center (MRTC) in Bamako, Mali and the National Institutes of Health (NIH) in the United

States. This protocol supports that research by ensuring a supply of blood samples from healthy Malian adults in order to

establish normal immunologic parameters for this population and to optimize research assays performed at the MRTC.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 - 55 years
* Resident of Kambila, Tieneguebougou or Kalifabougou
* Adequate venous access
* Willingness to allow blood samples to be stored and used for future studies of the immune response to malaria
* Ability to give informed consent and willingness to comply with study requirements and procedures

EXCLUSION CRITERIA:

* Anemia (hemoglobin less than 11 g/dL).
* Currently taking antimalarials, corticosteroids or other immunosuppressants.
* Underlying heart disease, bleeding disorder, or other conditions that in the judgment of the Principal Investigator (PI) could increase the risk to the volunteer.
* Fever greater than or equal to 37.5 degrees Celsius or evidence of an acute infection.
* Current pregnancy, as determined by urine dipstick test for pregnancy.
* Participation in another clinical protocol that requires the administration of an experimental vaccine or experimental treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults in a malaria endemic area in Mali
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Establishing immunological parameters | Before and during the 6-month malaria season
  Establishing immunological parameters in healthy malaria-exposed adults including phenotypic and functional measurements of dendritic cells, monocytes, NK cells, B cells and T cells

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Crompton, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- U Mali Faculty Med Pharmacy & Dentistry IRB #1, Bamako, Mali